CLINICAL TRIAL: NCT05829746
Title: PROSPECTIVE, MULTI-CENTER, OPEN-LABEL, SINGLE-ARM REGISTRATION TRIAL OF THE TUBRIDGE FOR THE TREATMENT OF WIDE-NECKED SMALL AND MEDIUM-SIZED INTRACRANIAL ANEURYSMS：PARAT MINI
Brief Title: PROSPECTIVE, MULTI-CENTER, OPEN-LABEL, SINGLE-ARM REGISTRATION TRIAL OF THE TUBRIDGE FOR THE TREATMENT OF WIDE-NECKED SMALL AND MEDIUM-SIZED INTRACRANIAL ANEURYSMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tubridge-2022-02-0A
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Brain Diseases; Aneurysm; Intracranial Aneurysm; Cardiovascular Diseases
MeSH Terms: conditions — Brain Diseases; Aneurysm; Intracranial Aneurysm; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Microport NeuroTech Tubridge flow-diverter Stent
  Interventions: Device: Tubridge

INTERVENTIONS:
Device: Tubridge — Intracranial stent for wide-necked aneurysms

SUMMARY:
A trial to evaluate the safety and efficacy of the Tubridge flow-diverter stent for the treatment of intracranial wide-necked, small to medium-sized aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-75 years;
* (2) Subjects with small to medium-sized aneurysms (aneurysm maximum diameter <10 mm) of the internal carotid artery or vertebral artery diagnosed by CTA, MRA or DSA angiography(including saccular aneurysms and recurrent saccular aneurysms) ;
* (3) Aneurysm neck ≥ 4 mm or aneurysm body to neck ratio < 2;
* (4) Parent artery diameter of 2.0 mm to 6.5 mm;
* (5) Subjects suitable for treatment with the Tubridge stent alone or in combination with coil;
* (6) The subject is willing to be followed up in accordance the protocol;
* (7) The subject or the subject's guardian understands the purpose of the trial, voluntarily to participate and sign the informed consent form.

Exclusion Criteria:

* (1) Aneurysm associated with AVM, MMD;
* (2) Ruptured aneurysms within 30 days;
* (3) Multiple aneurysms;
* (4) Subjects with severe stenosis (≥50% stenosis) or occlusion of the parent artery;
* (5) Aneurysms that have recurred after treatment with stents or stent-assisted coiling embolization
* (6) Subjects with morphology or lesions that may interfere with the use of device , including but not limited to: carotid artery entrapment, vasculitis, aortic entrapment, restricted vascular access (e.g., severe intracranial vascular tortuosity, severe intracranial vasospasm that does not respond to pharmacologic therapy, other anatomic or clinical lesions that prevent device access)
* (7) Subjects who are unsuitable for anesthesia or endovascular surgery, such as major diseases of the heart, lungs, liver, spleen, or kidneys, malignant tumors of the brain, severe active infections, disseminated intravascular coagulation, and a history of severe psychiatric disorders;
* (8) Subjects who have undergone major surgical procedures (e.g., implantation of internal fixation devices for fractures of the extremities, tumor resection, surgery on vital organs, etc.) within 30 days prior to signing the informed consent form or planned within 60 days after signing the informed consent form;
* (9) mRS score ≥ 3;
* (10) Subjects with a life expectancy of less than 12 months;
* (11) Subjects who have participated in other drug or medical device clinical trials prior to enrollment and have not met the study endpoint time frame;
* (12) Subjects who, in the judgment of the investigator, have poor adherence and are unable to complete the study as required;
* (13) Subjects with a suspected history of allergy to materials such as nickel-titanium, platinum, or platinum-iridium alloys;
* (14) Subjects who are unable to receive antiplatelet aggregation or anticoagulation therapy;
* (15) Subjects who have had or are likely to have a reaction to contrast agents so severe that they are unable to complete pre-treatment medication;
* (16) Women who are pregnant or breastfeeding;
* (17) Other conditions deemed by the investigator to be inappropriate for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete occlusion rate of aneurysms | 180±30 days
  The Raymond-Roy intracranial aneurysm occlusion classification was used to assess the rate of aneurysm occlusion postoperatively or at the time of primary endpoint assessment (12 months). Occlusion rates were reported as Class I: complete occlusion; Class II: residual neck; Class III: residual aneurysm.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided